CLINICAL TRIAL: NCT02448940
Title: The Effect of Supplementation With Species of Lactobacillus on Anthropometric Measurements, Body Composition, Appetite and Serum Lipid Profile in Overweight and Obese Adults
Brief Title: The Effect of Supplementation With Species of Lactobacillus on Anthropometric Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Urmia University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: umsu.rec.1393.74
Record Dates: First submitted 2015-05-06; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2014-06

CONDITIONS: Overweight and Obesity
Keywords: probiotics; Lactobacillus; obesity; body composition
MeSH Terms: conditions — Overweight; Obesity | interventions — Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Species of Lactobacillus (Experimental): 2 capsule/day of Lactofem Containing Species of Lactobacillus
  Interventions: Dietary Supplement: Species of Lactobacillus
- lactose (Placebo Comparator): 2 capsule/day Containing lactose
  Interventions: Dietary Supplement: lactose

INTERVENTIONS:
Dietary Supplement: Species of Lactobacillus — 2 capsule a day Lactofem probiotics containing Species of Lactobacillus
  Arms: Species of Lactobacillus
Dietary Supplement: lactose — 2 capsule a day containing lactose
  Arms: lactose

SUMMARY:
The investigators aimed to study the effect of supplementation with species of Lactobacillus on anthropometric measurements, body composition, appetite and serum lipid profile in overweight and obese adults

DETAILED DESCRIPTION:
The Objective of This Study was Evaluating the Effect of supplementation with Species of Lactobacillus on anthropometric measurements include weight, waist and hip circumference , body composition include body fat and muscle percent, appetite measured by visual analogues scale and serum lipid profile in overweight and obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* BMI more than 25 Kg/m2

Exclusion Criteria:

* taking drugs that could affect weight change, including anti-diabetic drugs, lipid lowering drugs
* endocrine,cardiovascular, thyroid, or chronic liver disease.
* had received surgery to reduce weight
* taking probiotics or antibiotics within one month
* Pregnancy or lactation or menopause
* A history of cancer
* Heart disease - cardiovascular, pulmonary, renal and diabetes
* A history of autoimmune disease
* Taking certain medications such as blood pressure control, statins, insulin sensitivity enhancers
* weight change over five percent within three months
* change in activity or diet habit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
weight change | Change from Baseline in body weight at 12 weeks

SECONDARY OUTCOMES:
defecation | Baseline,4 weeks, 8 weeks, 12 weeks
  Bristol stool scale (BBS)
blood pressure | Baseline,12 weeks
  include systolic and diastolic blood pressure
Anthropometric Measurement BMI | Baseline,4 weeks, 8 weeks, 12 weeks
  Body Mass Index (BMI) kg/m2
Anthropometric Measurement WC | Baseline,12 weeks
  waist circumference (WC) measures by "cm"
Anthropometric Measurement HC | Baseline,12 weeks
  hip circumference (HC) measures by "cm"
Appetite | Baseline,4 weeks, 8 weeks, 12 weeks
  numeric analogue Scale (NAS) mm
Anthropometric Measurement WHR | Baseline,12 weeks
  waist to hip ratio (WHR)
mid arm circumference Measurement | Baseline,12 weeks
Serum Lipid Profile | Baseline,12 weeks
skinfold thickness | Baseline,12 weeks
  triceps, biceps, supra iliac and subscapular skinfold
body fat percent | Baseline,12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Alizadeh, PhD, Principal Investigator — Department of Nutrition, School of Medicine, Urmia University of Medical Sciences
Locations (1):
- sardrood Clinic, Tabriz, Iran